CLINICAL TRIAL: NCT02490566
Title: Piloting Enhanced Pediatric Care for Children With Chronic Condition/Technology Trial
Brief Title: Enhanced Primary Care and Technology for Children With Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Verizon Wireless (Industry)
Responsible Party: Principal Investigator, Judy Schaechter, M.D., M.B.A., Chair of the Department of Pediatrics, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20140732
Record Dates: First submitted 2015-06-29; First posted 2015-07-07 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Overweight; Obesity; Asthma
Keywords: chronic condition; telehealth; nutrition; exercise
MeSH Terms: conditions — Overweight; Obesity; Asthma; Chronic Disease; Motor Activity | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Technology Arm (Experimental): Tablet computer with chronic disease apps will be given to patients. This tablet will also be used for follow-up visits done via video conferencing. Intervention: Telehealth.
  Interventions: Other: Telehealth

INTERVENTIONS:
Other: Telehealth — Tablet with chronic disease apps will be given to this group, apps will be focused on patient's condition. Follow-up visits will be conducted through video-conferencing.

SUMMARY:
Using technology alongside a pediatric chronic disease specialist and behavior specialist, the investigators are planning to help care for and coordinate the healthcare of children with chronic diseases, particularly childhood obesity, diabetes and asthma in Miami's most vulnerable communities. The University of (UM) Miller School of Medicine (MSOM) Pediatrics and TeleHealth departments propose to leverage information and communications technologies (ICT) in an innovative approach to improve the quality, access and efficiency of pediatric services for children and their families.

DETAILED DESCRIPTION:
Participants will be recruited from an outpatient clinic site with diagnoses of overweight, obesity or asthma.

There will be a total of 6 visits during the study at approximately 1 month intervals. During the first and last visits, pre- and post-intervention assessment points, quality of life, adherence to medical regimen, physical activity and dietary habits will be gathered. During the follow-up visits, only quality of life will be surveyed. At the initial visit, for overweight children, the patients will be assessed for their behaviors and attitudes regarding eating, physical activity, sedentary time and motivation. If the patient has asthma, the pediatrician will assess understanding of the disease.

Throughout the course of the study the chronic condition pediatrician and behavior specialist will see patients in a consult capacity for their chronic condition, but the patient will continue to see their regular pediatrician for primary care needs. At every visit the pediatrician will review changes since the last visit, and then provide education directed at overweight/obesity and/or asthma. The behavior health specialists will then work with the patients to develop a plan on how to follow their treatment plan and achieve healthy behaviors.

All of the participants will receive access to technology in the form of a tablet computer for the duration of the study. The tablets will be installed with software to help educate patients and their families about asthma and overweight/obesity and track progress in managing them. In addition, all follow-up visits except for the final one will be done using the tablets and a video-conferencing app.

For the first and last visits, all patients will be seen in-person in the clinic. All of the follow-up visits will be done via a video-conferencing app on the tablet computers.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive care at the Borinquen Clinic
* Aged five through 18, inclusive
* Diagnosis of asthma (requiring medication) or overweight (greater than or equal to 85% for age).
* Fluent in English or Spanish.
* Parents/Guardians must be fluent in English or Spanish.

Exclusion Criteria:

* None.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants compliant with supportive care visits | month 6
  Measure supportive care visits attended by participants

SECONDARY OUTCOMES:
Effect of telehealth on participants knowledge of their chronic condition | month 6
  Change in knowledge surveys given pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Schaechter, M.D., M.B.A., Principal Investigator — University of Miami
Locations (1):
- Borinquen Health Care Center, Miami, Florida, United States